CLINICAL TRIAL: NCT00860730
Title: PERCEVAL Pivotal Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corcym S.r.l (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V10801
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2019-01

CONDITIONS: Aortic Valve Replacement
Keywords: Aortic valve replacement; Aortic stenosis; Biological valve; Sutureless valve; Stented valve; Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Perceval S (Experimental)
  Interventions: Device: Aortic valve replacement with Perceval aortic heart valve

INTERVENTIONS:
Device: Aortic valve replacement with Perceval aortic heart valve — Replacement of diseased or malfunctioning native aortic valve via traditional surgery (open chest) with the Perceval S prosthesis

SUMMARY:
The clinical investigation is designed as a prospective and non-randomised study on a maximum of 150 patients. This study will be conducted at Investigational Centres in the European Community. A minimum number of 8 European Centres will be involved in the clinical investigation. A minimum of 15 patients will be enrolled at each Investigational Centre. The clinical follow-up requires evaluations at discharge (or 30 days if the patient is still hospitalized), 3-6 and 12 months following the procedure.The primary objective of this clinical investigation is to assess the performance of the Perceval S valve at 3-6 months after implantation in high surgical risk patients, who require a surgical intervention to replace the aortic valve.

DETAILED DESCRIPTION:
The design of the Perceval S prosthesis stems from the intention to offer an alternative to traditional flexible prostheses (stented and stentless biological valves) using conventional open-heart surgery. As a result of the sutureless implant procedure, in fact, patients could benefit from:

Reducing aortic clamp times, with subsequent overall reduction of surgical timing and therefore reduction in related risks; Avoiding to pass the stitches through the annulus and sutures knotting, with consequent less risk of tearing aortic annulus and wall, damaging the bundle of His, embolizing foreign material in the vascular system.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of 75 years or older;
* Subjects with aortic valve stenosis or steno-insufficiency;
* Subjects at high surgical risk and candidates for aortic valve replacement with a biological prosthesis;
* Subjects in NYHA functional classes III and IV with the Logistic EuroSCORE greater than 5%.
* Subjects who have agreed to participation in the clinical evaluation and who have signed the informed consent;
* Subjects who are willing to undergo all the medical follow-ups and echocardiographic examinations and laboratory tests that form part of this present protocol.

Exclusion Criteria:

* Subjects involved in any other clinical study for drugs or devices;
* Subjects who have previously undergone implantation with the Perceval S prosthesis being assessed;
* Subjects with previous implantation of valve prostheses or annuloplasty ring in mitral position;
* Subjects requiring simultaneous procedures, apart from septal myectomy and/or coronary by-pass;
* Subjects with aneurysmal dilation or dissection of the ascending aortic wall needing surgical correction;
* Subjects needing non elective intervention;
* Subjects with aortic annulus (after procedure for decalcification) of dimensions such that the implantation of a valve of size 21 or 23 mm is not possible (direct intra-operative measurement with sizer), in accordance with the indications reported in the Investigator's Brochure;
* Subjects with active endocarditis;
* Subjects with active myocarditis;
* Subjects with any anomaly of the coronary ostia determined through pre-operative coronary angiogram or during intervention itself;
* Subjects with congenital bicuspid aortic valve;
* Subjects with aortic root enlargement, where the ratio between observed and expected diameters (calculated as a function of age and patient body surface area) is > 1.3;
* Subjects with aortic root enlargement, where the ratio between the diameter of the sino-tubular junction and the annulus diameter is > 1.3;
* Subjects with myocardial infarct < =90 days;
* Subjects with known hypersensitivity to nickel alloys.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety of the Perceval S prosthesis in terms of percentage incidence of mortality and morbidity at 3-6 months after implant | 6 months

SECONDARY OUTCOMES:
Assessment of mortality and morbidity rates at discharge (or 30 days if the patient is still hospitalized) and 12 months after implant | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Axel Haverich, Prof, Principal Investigator — Hannover Medizinische Hochschule
Locations (9):
- UZ Leuven, Leuven, Belgium
- France (4):
  - CHRU de Lille, Lille
  - Hopital Guillaume et René Laennec, Nantes
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Cardiologique du Haut-Lévêque, Pessac
- Germany (3):
  - Ruhr Universität Bochum, Bochum
  - Westdeutsches Herzzentrum, Essen
  - Medizinische Hochschule Hannover, Hanover
- Inselspital Bern, Bern, Switzerland

REFERENCES:
- See also: Website — http://www.sorin.com